CLINICAL TRIAL: NCT03719638
Title: Comparison of Two Blades of Videolaryngoscope in Simulated Difficult Airway in Children, a Randomized Controlled Trial
Brief Title: Comparison of Two Blades of Videolaryngoscope in Simulated Difficult Airway in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Alparslan Kus, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2018-154
Record Dates: First submitted 2018-10-20; First posted 2018-10-25 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Intubation;Difficult
Keywords: D-Blade; Macintosh videolaryngoscope blade; Simulated difficult intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-blade group (Active Comparator): Intubation will be done using D-blade of videolaryngoscope in a simulated difficult airway Difficult airway will be simulated with collar.
  Interventions: Device: D-blade of videolaryngoscope; Other: simulated difficult airway
- Macintosh group (Active Comparator): Intubation will be done using Macintosh videolaryngoscope in a simulated difficult airway Difficult airway will be simulated with collar.
  Interventions: Other: simulated difficult airway; Device: Macintosh videolaryngoscope

INTERVENTIONS:
Device: D-blade of videolaryngoscope — intubation will be done using d-blade of videolaryngoscope
  Arms: D-blade group
Other: simulated difficult airway — extension of head will be limited by using collar.
Device: Macintosh videolaryngoscope — intubation will be done using macintosh videolaryngoscope
  Arms: Macintosh group

SUMMARY:
Airway management and tracheal intubation are routinely performed in paediatric anaesthesia and yet are associated with preventable adverse events. The D-blade of videolaryngoscope is preferred in difficult intubation with a more curved blade then the Macintosh videolaryngoscope blade, which may be more useful in difficult intubation. The aim of the study is to compare the D-blade of videolaryngoscope with Macintosh videolaryngoscope blade.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Undergoing elective surgeries
* Age between 1-5 years

Exclusion Criteria:

* Anticipated difficult intubation
* Pulmonery diseases
* >III ASA scores

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
intubation time | time between handling videolaryngoscope and inserting endotracheal tube
  Time of endotracheal intubation will be recorded.

SECONDARY OUTCOMES:
Cormack and Lehane score | During the intubation
  Cormack and Lehane scores from 1 to 4 where 1 is the best and 4 is the worst score for laryngoscopy view will be recorded for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Kus, MD, Principal Investigator — Kocaeli University School of Medicine
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No